CLINICAL TRIAL: NCT05962333
Title: Assess Effect and Safety of Intra-arterial Autologous Mesoangioblast Administration to the Upper Arm of m.3243A>G Mutation Carriers
Brief Title: Effect and Safety MABs Administration m.3243A>G Mutation Carriers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL82815.000.22
Record Dates: First submitted 2023-05-23; First posted 2023-07-27 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Mitochondrial Myopathies
Keywords: m.3243A>G; mesoangioblasts
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Intervention Model Description: Intra-subjected controlled clinical study. Treatment is performed in left arm of the subjects and right arm (no intervention), measurements are performed before the first and after the last administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-arterial delivery of autologous MABs (Experimental): Autologous MABs will be injected three times in left arm to treat biceps brachii muscle
  Interventions: Biological: Intra-arterial delivery of autologous MABs

INTERVENTIONS:
Biological: Intra-arterial delivery of autologous MABs — three times intra-arterial administration of autologous mesoangioblasts in biceps brachii of the left arm at 4-6 week interval

SUMMARY:
The first primary objective is to assess the effect of three intra-arterial administrations of autologous mesoangioblasts (MABs) with respect to improving muscle strength and reduce fatigue of the treated biceps brachii (BB) compared to the untreated BB.

The second primary objective is safety of three intra-arterial administrations of autologous MABs, which the investigators will assess by monitoring (serious) adverse events ((S)AEs), blood flow in left arm pre- and post-intervention, and neurological vital signs during 8h post-intervention observation in the hospital.

Secondary objectives are to assess changes in muscle mass of the treated and untreated BB muscle, and microscopic changes and m.3243A>G mutation load at tissue level in treated biceps brachii (BB) muscle at baseline and after treatment.

Up to 20 adult m.3243A>G patients will undergo a ~30mg m. biceps brachii muscle biopsy at visit 1. The first six eligible patients will enroll the clinical study based on their m.3243A>G mutation load in skeletal muscle (50-90%) and mesoangioblasts (<10%), and on a decreased BB muscle strength and increased fatigue.

These 6 selected patients will visit the Maastricht University Medical Center for 8 additional times. From each patient, during visit 2 till 9:

* BB muscle biopsies of the left arm will be collected (1x ~130 mg at visit 2 and 1x ~30mg at visit 9)
* MRI of the BB muscles in both arms will be performed (visit 2 and 9).
* Autologous MABs will be injected into the left arm via axillary artery delivery. Angiography will be performed before and after infusion to assess vascular obstructions, and the participant will be monitored in the hospital for 8 hours (visit 4,6,8).
* Tc99m macroaggregated albumin (MAA) is infused to quantify blood flow to the BB muscle (visit 4).
* A bout of maximal eccentric exercise of BB muscles on both sides will be executed at visit 3, 5 and 7.
* BB muscle strength will be assessed using a Biodex dynamometer (visit 3-9)
* venous blood samples will be taken for assessing muscle damage and inflammation markers (visit 3-9), kidney functioning, coagulation and viral screening (visit 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age: 18-64
* Sex: male/female
* Patients with the m.3243A>G mutation load of 50%-90% determined in skeletal muscle or derived from age-corrected calculation of blood m.3243A>G mutation load

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Use of dabigatran, apixaban, edoxaban or rivaroxaban (DOACs) as anti-coagulants
* Have a weekly alcohol intake of ≥ 35 units (men) or ≥ 24 units (women)
* Current history of drug abuse
* Deficient immune system or autoimmune disease
* Significant concurrent illness
* Ongoing participation in other clinical trials with intervention
* Pregnant or lactating women
* Psychiatric or other disorders likely to impact on informed consent
* Patients unable and/or unwilling to comply with treatment and study instructions
* A history of strokes with signs of extra-pyramidal or pyramidal syndrome
* Allergy for contrast fluid
* Peripheral signs of ischemia or vasculopathy
* Claustrophobia
* Metal implants
* Any other factor that in the opinion of the investigator excludes the patient from the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess blood flow in left arm following i.a. arterial delivery of autologous MABs | before and directly after each administration in week 1,5 and 10
  Assess blood flow in left arm using digital subtraction angiography (DSA) before and directly after MABs administration in week 1, 5 and 10.
Assess (serious) adverse events following 3 i.a. deliveries of autologous MABs | 15 weeks
  Assessment of (serious) adverse events
Assess temperature following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Temperature will be checked 0,1,2,3,4,6 and 8 hours after administration in week 1,5 and 10.
Assess oxygen saturation following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Oxygen saturation will be checked 0,1,2,3,4,6 and 8 hours after administration in week 1,5 and 10.
Muscle strength arm following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Using Medical Research Council (MRC) scale for muscle strength, muscle strength of left arm will be assessed 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10. MRC scale ranges from 0 (no visible contraction) to 5 (normal)).
Assess breathing frequency following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Breathing frequency will be checked 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10.
Assess vital signs following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Heart rate will be checked 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10.
Assess systolic and diastolic blood pressure following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Systolic and Diastolic blood pressure will be checked 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10.
Assess Glasgow Coma scale (GCS) score following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  Glasgow Coma Scale (GCS) score will be determined 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10. GCS score ranges from 3 to 15, 3 being the worst and 15 being the best score.
Assess if pupil size is symmetrical in both eyes following 3 i.a. deliveries of autologous MABs | 0, 1,2,3,4,6 and 8 hours after each administration.
  Pupil size of both eyes will be assessed 0,1,2,3,4,6 and 8 hours after administration in week 1, 5 and 10. If pupil size is not equal, this can indicate disease or trauma.
Assess pupil reaction following 3 i.a. deliveries of autologous MABs | 0,1,2,3,4,6 and 8 hours after each administration.
  To assess brain functioning, reaction of pupils to light will be determined 0,1,2,3,4,6 and 8 hours after administration. Upon light, both pupils should become smaller in week 1, 5 and 10. No reaction or only reaction in one eye can indicate nerve damage.
Assess changes in muscle strength of biceps brachii muscle in both arms at baseline and 4-6 weeks after third i.a. delivery of autologous MABs in left arm, which is 12-16 weeks after baseline measurements. | baseline and 15 weeks after 1st administration
  Determine maximum muscle force generating capacity (peak torque N/m) of the biceps brachii muscle in both arms using Biodex dynamometer measurements. Measurements will be performed in left (intervention) and right (no intervention) biceps brachii muscle using Biodex dynamometer measurements at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.
Assess changes in muscle fatigue of biceps brachii muscle in both arms at baseline and 4-6 weeks after third i.a. delivery of autologous MABs in left arm, which is 12-16 weeks after baseline measurements. | baseline and 15 weeks after 1st administration
  Asses changes in muscle fatigue by measuring percentage decrease in maximum muscle force generating capacity (peak torque N/m) between first and sixth repetition. Measurements will be performed in left (intervention) and right (no intervention) biceps brachii muscle using Biodex dynamometer measurements at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.

SECONDARY OUTCOMES:
Assess changes in muscle volume biceps brachii muscles of both arms following 3 i.a. deliveries of autologous MABs in left arm. | baseline and 15 weeks after 1st administration
  MRI T3 analysis to assess changes in muscle volume in both arms at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.
Assess formation of new muscle fibers following 3 i.a. deliveries of autologous MABs | baseline and 15 weeks after 1st administration
  Perform embryonic myosin heavy chain (MHC)+ immunostaining to assess percentage of new / regenerating muscle fibers in muscle biopsies collected at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.
Mitochondrial mutation load and functioning following 3 i.a. deliveries of autologous MABs | baseline and 15 weeks after 1st administration
  Assess changes in m.3243A>G mutation load in new/regenerating muscle fibers compared to existing muscle fibers isolated via laser microdissection from muscle biopsies left arm collected at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.
Mitochondrial functioning following 3 i.a. deliveries of autologous MABs in left arm. | baseline and 15 weeks after 1st administration
  Assess changes in mitochondrial functioning by performing Cytochrome C Oxidase / Succinate Dehydrogenase (COX/SDH) staining in muscle biopsies from left arm collected at baseline and 5 weeks after the third autologous MABs administration, which is 15 weeks after baseline measurements.

OTHER OUTCOMES:
Assess creatine kinase level in blood plasma as marker for muscle damage following 3 i.a. deliveries of autologous MABs | 0 and 8 hours after each administration.
  Assess creatine kinase (CK) in blood plasma following eccentric exercise prior and 8 hours after administration in week 1,5 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Janneke Hoeijmakers, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Tienen F, Zelissen R, Timmer E, van Gisbergen M, Lindsey P, Quattrocelli M, Sampaolesi M, Mulder-den Hartog E, de Coo I, Smeets H. Healthy, mtDNA-mutation free mesoangioblasts from mtDNA patients qualify for autologous therapy. Stem Cell Res Ther. 2019 Dec 21;10(1):405. doi: 10.1186/s13287-019-1510-8. PMID 31864395
- See also: website Generate Your Muscle (GYM) project — http://www.generateyourmuscle.com